CLINICAL TRIAL: NCT01732146
Title: Phase III Study of Efficacy of High Dose Erythropoietin to Prevent Hypoxic-ischemic Encephalopathy Sequelae in Term Newborn
Brief Title: Efficacy of Erythropoietin to Improve Survival and Neurological Outcome in Hypoxic Ischemic Encephalopathy
Acronym: Neurepo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P110111; 2012-001417-17 (EudraCT Number)
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Hypoxic Ischemic Encephalopathy; Term neonate; Neuroprotection; erythropoietin
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Parturition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin beta (Active Comparator): 1000 to 1500 U/kg/dose X 3 every 24 hours
  Interventions: Drug: erythropoietin Beta
- Placebo (Placebo Comparator): 0.2 ml saline solution X 3 given every 24 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: erythropoietin Beta — erythropoietin intravenous injection (5000 U/ 0.3 ml)1000 to 1500 U/kg/dose X 3 given every 24 hours with the first dose within 12 hours of delivery
  Arms: Erythropoietin beta
Drug: Placebo
  Other Names: 0.2 ml saline solution X 3 given every 24 hours with the first dose within 12 hours of delivery
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of high dose Erythropoietin to improve survival and neurologic outcome in asphyxiated term newborn undergoing cooling.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy remains the main cause of death or long term neurologic impairments in neonates. Yet, therapies for birth asphyxia are currently limited. Hypothermia when applied within 6 hours after birth demonstrate partial improvement in outcome of newborns specially those with moderate form. Erythropoietin and its receptors are upregulated after brain injury in ischemic conditions. Systemically administered erythropoietin is neuroprotective in animal models of birth asphyxia. To date, one study demonstrate improvement neurologic outcome in asphyxiated term newborn under erythropoietin treatment but no reports evaluating beneficial of erythropoietin associated with cooling. This is a large randomised controlled trial to evaluate the efficacy of high dose erythropoietin on outcome at two years of asphyxiated term newborns undergoing cooling.

ELIGIBILITY:
Inclusion Criteria:

* Term or near-term newborn (> = 36 weeks gestational age)
* Moderate to severe encephalopathy
* undergoing moderate controlled hypothermia started within 6 hours after delivery : rectal or esophageal temperature maintained at 33.5 ° C + / - 0.5 ° C before H6
* Beneficiary of social security plan
* Informed consent parental authority

Exclusion Criteria:

* Impossibility of getting controlled hypothermia before H6
* Infant older than 12 hours of age
* Chromosomal or significant congenital abnormality
* Predictable surgery in the first 3 days of life
* Uncontrolled collapse
* Haemorrhagic syndrome unchecked
* Head trauma with or without skull fracture

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2013-03-28 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Survival without neurologic sequelae | at 24 months

SECONDARY OUTCOMES:
Mortality rates | Within 24 months
  number of dead patients
Rate of moderate and severe sequelae | at 24 months
  Mental Developmental index (Brunet Lezine Test), motor, visual and hearing impairment
Aspect of brain lesions on MRI | at day 6 and day 12 after birth
  Brain MRI performed between day 6 and day 12 after birth
Tolerance of treatment | at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Patkai, MD, PhD, Principal Investigator — Cochin Hospital
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Background] Zhu C, Kang W, Xu F, Cheng X, Zhang Z, Jia L, Ji L, Guo X, Xiong H, Simbruner G, Blomgren K, Wang X. Erythropoietin improved neurologic outcomes in newborns with hypoxic-ischemic encephalopathy. Pediatrics. 2009 Aug;124(2):e218-26. doi: 10.1542/peds.2008-3553. Epub 2009 Jul 27. PMID 19651565
- [Background] Goodarzi MO, Carmina E, Azziz R. DHEA, DHEAS and PCOS. J Steroid Biochem Mol Biol. 2015 Jan;145:213-25. doi: 10.1016/j.jsbmb.2014.06.003. Epub 2014 Jul 5. PMID 25008465